CLINICAL TRIAL: NCT04485065
Title: A Phase Ib Study Evaluating the Safety and Efficacy of IBI188 in Combination With Azacitidine in Subjects With Newly Diagnosed Higher Risk Myelodysplastic Syndrome
Brief Title: Safety and Efficacy of IBI188 With Azacitidine in Subjects With Newly Diagnosed Higher Risk MDS
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Suspended for changes in development strategy
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI188C301
Record Dates: First submitted 2020-07-21; First posted 2020-07-24 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Myelodysplastic Syndromes
Keywords: MDS
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IBI188+azacitidine (Experimental)
  Interventions: Drug: IBI188+azacitidine

INTERVENTIONS:
Drug: IBI188+azacitidine — Escalating and maintenance dose of IBI188 will be administered 30mg/kg, IV(intravenous infusion),Q4W
  Drug:Azacitidine Azacitidine will be administered daily for 7 days, IH, Q4W

SUMMARY:
The study is to evaluate safety and efficacy of IBI188 in combination with azacitidine (AZA) as a first-line treatment in subjects with newly diagnosed higher risk myelodysplastic syndrome

ELIGIBILITY:
Inclusion Criteria:

1. MDS subjects with higher risk;
2. Age ≥ 18 years old;
3. Eastern Cooperative Oncology Group score of 0~1;
4. Not suitable for or refuse to receive HSCT;
5. Newly diagnosed MDS subjects;
6. Adequate organ function;
7. Subjects should take effective contraceptive measures
8. Must sign the Informed Consent Form (ICF), and be able to follow all study procedures.

Exclusion Criteria:

1. Subject who has transformed from MDS to AML.
2. Therapy-related MDS (t-MDS), myeloproliferative neoplasm (MPN)- transformed MDS,MDS/MPN.
3. MDS subjects with lower risk.
4. Subjects who have received chemotherapy.
5. Prior exposure to any anti-CD47 or anti-SIRPα agents.
6. Subjects participating in another interventional clinical study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-09-30 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-08-20 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | 24 months
  To evaluate the safety and tolerability of IBI188 combined with Azacitidine (AZA) in first-line treatment of Myelodysplastic syndrome (MDS)
Complete response rate (CR) and duration of complete response (DoCR) | 24 months
  Complete response rate (CR) and duration of complete response (DoCR) in high-risk MDS subjects with IBI188 combined with AZA as first-line therapy evaluated by the central laboratory.

SECONDARY OUTCOMES:
Complete response rate (CR) and duration of complete response (DoCR) | 24 months
  Complete response rate (CR) and duration of complete response (DoCR) in high-risk MDS subjects with IBI188 combined with AZA as first-line therapy evaluated by the investigators;

CONTACTS AND LOCATIONS:
Locations (1):
- Blood Diseases Hospital Chinese Academy Of Medical Science, Tianjin, China